CLINICAL TRIAL: NCT01862016
Title: Early Spontaneous Breathing in Acute Respiratory Distress Syndrome
Acronym: BiRDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2009-04; 2012-A00551-42 (Other: IDRCB number (ANSM))
Record Dates: First submitted 2013-05-17; First posted 2013-05-24 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; APRV ventilatory mode; Spontaneous breathing; Intensive Care Unit
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAC mode, Controlled ventilation (Active Comparator): From randomization, patients are put under controlled ventilation with specific settings
  Interventions: Biological: arterial blood gas measurement each morning
- APRV mode, Spontaneous breathing (Experimental): During 1 to 3 hours after randomization, patients are put under controlled ventilation with specific settings for baseline data. After that, they are placed under APRV mode with specific settings
  Interventions: Procedure: APRV; Biological: arterial blood gas measurement each morning

INTERVENTIONS:
Procedure: APRV — Pressure ventilation mode allowing early spontaneous breathing
  Arms: APRV mode, Spontaneous breathing
Biological: arterial blood gas measurement each morning

SUMMARY:
The care of acute respiratory distress syndrome (ARDS) has been significantly improved by learning from experimental and physiological research works and by a series of randomized controlled trials. The mortality of this syndrome remains however high. Numerous experimental and clinical works demonstrated that a ventilatory mode authorizing the patient to make, from the acute phase, spontaneous breathing cycles superimposed on assistance delivered by the ventilator (BIPAP-APRV mode) allowed to improve gas exchanges and hemodynamic tolerance of the ventilation while reducing the need for sedative drugs. This ventilatory mode could also reduce the risk of diaphragmatic dysfunction induced by ventilation. Consequently, our hypothesis is that this ventilatory mode could allow a reduction of mortality in ARDS patients.

The aim of this multicenter, prospective, randomized, controlled, open study is to compare the effects of two ventilatory strategies on the mortality of ARDS patients and placed under mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Within 1 week of a known clinical insult or new or worsening respiratory symptoms
* Intubation and mechanical ventilation
* Bilateral opacities - not fully explained by effusions, lobar/lung collapse, or nodules lung
* Report PaO2 / FiO2 ≤ 200 mmHg with a PEP of at least 5 cmH2O
* Respiratory failure not fully explained by cardiac failure or fluid overload
* Criteria 1, 2 and 3 presents jointly for less than 48 hours
* Consent to participate obtained either from the patient himself or from a relative.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Predictable duration of the mechanical ventilation on endotracheal tube lower than 48 hours
* Patient being in period of exclusion further to the participation in another biomedical study
* intracranial hypertension (suspected or confirmed)
* known or suspected COPD
* Chronic respiratory failure treated by long-term oxygen and / or long-term respiratory support
* Morbid obesity defined as weight greater than 1 kg / cm
* Sickle Cell Disease
* Marrow recent transplant, post-chemotherapy aplasia
* Widened burns (> 30% body surface area)
* Severe hepatic cirrhosis (Child-Pugh C)
* Pneumothorax (drained or not)
* Treatment with extracorporeal support (ECMO)
* Decision of active therapeutic limitation
* Unavailability of the model of respirator that must be used in the study
* Failure to obtain a consent by persons authorized to do so.
* Patient under law protection.
* Person non-beneficiary of a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
all cause hospital mortality | hospital discharge
  participants will be followed for the duration of hospital stay, until day 60 maximum.

SECONDARY OUTCOMES:
all causes mortality | Day 28
number of days alive without mechanical ventilation | day 28
number of days alive without organ failure | day 28
number of patients with refractory hypoxemia | day 7
number of patients requiring adjuvant treatment of hypoxemia | day 7
number of days alive without sedation | Day 28
total amount of sedative drugs | between baseline and day 7
amount of sedative drugs received daily living | between baseline and day 7
number of days alive without vasoactive drugs | day 28
total amount of vasoactive drugs | between baseline and day 7
amount of vasoactive drugs received daily living | between baseline and day 7
Number of patients with a pneumothorax | day 28
Duration of mechanical ventilation | day 60
Duration of stay in ICU | day 60
Changes in serum levels of proinflammatory cytokines | Hour 1 and Hour 48

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Intensive Care Unit, University Hospital of Angers, Angers, France